CLINICAL TRIAL: NCT00002818
Title: Phase I and Clinical Pharmacokinetic De-Escalation Study of 2'-Deoxycitidine Administered as a Continuous Infusion in Conjunction With a Continuous Infusion of High-Dose ARA-C in Patients With Refractory Acute Myelogenous Leukemia
Brief Title: High-Dose Cytarabine Plus Deoxycytidine in Treating With Acute Myelogenous Leukemia or Other Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000064976; P30CA016059 (NIH); MCV-MCC-9409-2CC (Registry Identifier: ClinicalTrials.gov); VCU-FDR000637 (Other: Food and Drug Administration); NCI-V96-0966 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2000-08-03; First posted 2004-04-22 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Drug/Agent Toxicity by Tissue/Organ; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm
Keywords: recurrent adult Hodgkin lymphoma; refractory multiple myeloma; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; drug/agent toxicity by tissue/organ; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Hodgkin Disease; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Blast Crisis; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Cytarabine; Deoxycytidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: cytarabine
Drug: deoxycytidine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Deoxycytidine may protect patients from the side effects of high-dose cytarabine.

PURPOSE: Phase I trial to study the effectiveness of high-dose cytarabine given with deoxycytidine in treating patients who have refractory acute myelogenous leukemia or other lymphoma or leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Estimate the lowest dose of deoxycytidine (dC) that can be given as a host protective agent in conjunction with high dose cytarabine (HD ARA-C) in patients with refractory acute myelogenous leukemia or other hematologic malignancies. II. Determine the maximum tolerated dose and dose-limiting toxic effects of HD ARA-C/dC in these patients. III. Characterize the pharmacokinetics of continuously administered HD ARA-C/dC in these patients. IV. Characterize, when possible, the pharmacodynamics of HD ARA-C, dC, and their metabolites in blasts obtained from leukemic patients participating in this trial. V. Recommend the lowest possible dose of dC that can be given in combination with HD ARA-C in future phase II trials.

OUTLINE: This is a dose escalation study. Patients receive deoxycytidine IV over 120 hours. Beginning 12 hours after initiation of deoxycytidine, patients receive high dose cytarabine IV over 96 hours. Patients achieving complete response receive no further therapy. Patients achieving partial response or initial complete response and subsequent relapse receive an additional course of therapy. Cohorts of 3-6 patients receive escalating doses of deoxycytidine and high dose cytarabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicities.

PROJECTED ACCRUAL: Approximately 24-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: One of the following histologically documented hematologic malignancies: Acute myelogenous leukemia Failed or relapsed following conventional dose chemotherapy (e.g., doxorubicin, cytarabine) or high dose cytarabine (HD ARA-C) Chronic myelogenous leukemia in blast crisis that has failed at least 1 conventional antileukemic regimen Acute lymphoblastic leukemia (ALL) that is relapsed following or initially refractory to conventional therapy Failed at least 1 salvage regimen for ALL Disease refractory to conventional HD ARA-C allowed Primarily refractory or relapsed Hodgkin's or non-Hodgkin's lymphoma Failed at least 1 conventional second or third generation regimen (e.g., ProMACE-CytaBOM) Refractory multiple myeloma Not eligible for protocols of higher priority and no alternative forms of therapy available that offer a reasonable chance of palliation or cure

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 50-100% Life expectancy: At least 8 weeks Hematopoietic: Not specified Hepatic: Bilirubin less than 3 mg/dL Renal: Creatinine clearance at least 40 mL/min Pulmonary: Pulse oximetry greater than 88% in patients with a history of pulmonary disease Other: No major concurrent disease that renders patient a poor medical risk No uncontrolled infection Disease related fever allowed at investigator's discretion No mental incapacity that precludes informed consent No incarcerated patients Not pregnant Effective contraception required of fertile women

PRIOR CONCURRENT THERAPY: Not specified Biologic therapy: Not specified Chemotherapy: At least 3 weeks since prior chemotherapy (24 hours since hydroxyurea) and recovered Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy to 30% or more of bone marrow At least 4 weeks since prior radiotherapy and recovered Surgery: Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 1995-02; Primary Completion 2001-02 (Actual); Study Completion 2001-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Grant, MD, Study Chair — Massey Cancer Center
Locations (1):
- Massey Cancer Center, Richmond, Virginia, United States